CLINICAL TRIAL: NCT03013660
Title: Supporting Mothers of Preterm Infants: A Randomized Controlled Trial
Brief Title: Supporting Mothers of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB15-3993; NCT02953795 (obsolete NCT alias)
Record Dates: First submitted 2016-11-04; First posted 2017-01-06 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: PreTerm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison (No Intervention): Participants will be provided with standard information about the benefits of STSC and breastfeeding and will be encouraged to come into the NICU every day for at least 1 hour of STSC. To facilitate increased let down of breast milk, all participants will be provided a hospital grade breast pump free of charge during the stay of their babies in the NICU and assistance will be provided to the mothers in procuring a Medicaid covered breast pump to keep when the baby leaves the NICU. The hospital grade breast pump will be provided to her as soon as she enrolls into the study and will remain with her until her baby is discharged or transferred.
- Treatment: Limited Financial Support (Experimental): Subjects randomized to this arm will be contacted to be informed that they are eligible to receive a weekly financial transfer to help them spend more time with their baby at the NICU. The intervention participants will be eligible to receive this transfer every 7 days, starting on the day of enrollment. The participants selected for the intervention arm will be asked not to discuss the payment with any other study participants (such as the members of any other families they may see at the NICU) or other health care staff at the NICU. Participants will also receive everything that the Comparison group receives.
  Interventions: Other: Limited Financial Support

INTERVENTIONS:
Other: Limited Financial Support — Subjects randomized to this arm will be contacted to be informed that they are eligible to receive a weekly financial transfer to help them spend more time with their baby at the NICU. The intervention participants will be eligible to receive this transfer every 7 days, starting on the day of enrollment.
  Arms: Treatment: Limited Financial Support

SUMMARY:
Preterm birth is the leading contributor to mortality among children younger than 5 years. One effective and inexpensive intervention is providing skin-to-skin care (STSC) whereby the mother of a preterm baby provides skin-to-skin contact to the newborn for at least a few hours, ideally every day. This intervention can make breastfeeding easier and can improve the health and development of the baby.

Unfortunately, despite the large health benefits, mothers in low-resource communities are often unable to practice STSC due to a range of institutional and economic barriers. STSC requires substantial time and financial commitments from mothers; they must travel from home each day to the hospital to engage in STSC and provide expressed breast milk. Low-income women with access only to limited federally provided unpaid family leave may have to choose between returning to work while their baby is in the NICU and being able to stay at home with their newborn after discharge from the NICU. Families of preterm infants also face direct financial costs of practicing STSC and breastfeeding (such as fees for parking and childcare for older children).

This trial aims to examine the impact of providing additional support to low-income mothers of babies born preterm in 2 hospitals in Massachusetts to help them provide STSC. Half of the participants will be randomized to receive an additional financial support intervention while their infant is in the NICU. The study will examine how this intervention impacts mothers' health behavior while their child is in the NICU and up to three months after.

Most of the current and past policy efforts to increase STSC have focused on the delivery of STSC at hospitals, focusing on supply-side related challenges such as the lack of trained and informed staff. However, interventions that focus exclusively on hospitals are unlikely to be sufficient for low-income women if there are significant opportunity costs or transportation costs to simply being present at the hospital. This study aims to provide more evidence to determine whether removing these financial barriers has the potential to mitigate the poor outcomes of preterm babies born to lower socioeconomic status households.

ELIGIBILITY:
Inclusion Criteria:

1. mothers who gave (preterm) birth at the study hospitals as well mothers who gave birth elsewhere (e.g. at a hospital without a high-level NICU) but whose babies were immediately transferred to the study hospitals for preterm care after birth.
2. mothers of children born between 30 and 36 weeks of gestation without any major complications requiring additional or special medical care for mother and child

Exclusion Criteria:

1. under the age of 18 years
2. not currently covered by Medicaid
3. unable to speak or understand English or Spanish
4. not residents of the state of Massachusetts
5. any of the following complications: HIV infection, active tuberculosis, are undergoing radiation therapy, recent breast surgery, indications of illicit drug use currently or during pregnancy (from meconium or cord sample, or urine test), or other contraindications for breastfeeding; or their baby has congenital, surgical, or cardiac anomalies. Note that enrolled women who are identified as using illicit drugs after enrollment will be removed from the study per hospital protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-07-05 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Proportion of days mothers practice STSC | Captured in hospital records during the first 1-3 weeks after enrollment
  Number of days enrolled mothers practice STSC divided by the total number of days their infant is stable in the NICU (count starts after enrollment)

SECONDARY OUTCOMES:
Exclusive breastfeeding duration | Self-reported after 3 months
  Mean weeks of exclusive breastfeeding duration among enrolled mothers
Change in head circumference | Head circumference measured at birth (time 0) and after 3 months
  Difference between head circumference z-score at birth and at 3 months post-discharge
General infant development composite score (based on 5 age-appropriate milestones) | Reported by mother at 3 month survey
  Infant development composite score as measured by 5 age-appropriate motor, communication, and socioemotional milestones
Mental/emotional wellbeing of mother | Self-reported after 3 months
  Mental/emotional wellbeing score of enrolled mothers based on Edinburgh Scale of Postpartum Depression
Mother-infant attachment | Self-reported after 3 months
  Attachment score between enrolled mothers and their preterm infant based on Postpartum Bonding Questionnaire
Readmissions | Self-reported after 3 months
  Fraction of infants who were readmitted to the hospital post-discharge
Cost and cost-effectiveness | Within 3 months of discharge
  Total cost of infant's care, including both hospital and out-of-pocket spending
Any breastfeeding at 3mo | Self-reported after 3 months
  Fraction of mothers still breastfeeding (does not need to be exclusive) their infants at 3 months
Breastfeeding initiation | Captured in hospital records during first 1-3 weeks after enrollment
  Fraction of mothers who ever begin breastfeeding
Duration of NICU stay | Captured in hospital records during the first 1-3 weeks after enrollment
  Number of days infants stay in the NICU before discharge
Change in weight-for-age z-score | Change between measurement at birth (time 0) and after 3 months after discharge
  Difference between birthweight z-score and weight-for-(corrected)-age z-score of infant at 3mo

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts

IPD SHARING:
Plan to Share IPD: No